CLINICAL TRIAL: NCT06116474
Title: Effect Of 8-Week Online Fitness Intervention on Muscle Strength, Flexibility, Body Composition and Physical-Self Perception
Brief Title: Effect Of 8-Week Online Fitness Intervention Health Related Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Technical University (Other)
Responsible Party: Principal Investigator, Gunay yildizer, Associated Professor, Eskisehir Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EkisehirTU-SBF-GY-01
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Sedentary Behavior; Physical Inactivity; Body Image
Keywords: Exercise; Leisure Activities
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web based intervention group (Experimental): The web-based intervention group participated in an 8-week exercise program, which consisted of three sessions per week, each lasting approximately 20 to 35 minutes.
  Interventions: Behavioral: Web-Based Physical Fitness Intervention
- Control Group (No Intervention): The control group did not engage in any prescribed exercise protocol.

INTERVENTIONS:
Behavioral: Web-Based Physical Fitness Intervention — The exercise program has been designed according to the progressive overload method. Therefore, the volume of the exercise program increased as the weeks progressed. Exercise videos were uploaded to YouTube on Mondays, Wednesdays and Fridays send to participants via a message group to follow the program. The videos featured the experts' explanations of the movements for each exercise.. The equipment that the participants should use in the training sessions was selected from the materials available at home (eg., use of water bottles instead of weight dumbbells). The exercise sessions is divided into 3 parts: warm-up (2-4 min. average), main part (14-19 min. average), cool-down (3-5 min. average). The warm-up includes movements to increase the heart rate and warm up the muscles to be worked on for that session. The main part of the exercise program also included rest breaks when the participants were asked to move and stretch.
  Arms: Web based intervention group

SUMMARY:
The purpose of this study is to investigate the effectiveness of 8-week online delivered exercise program on actual and perceived physical fitness components.

DETAILED DESCRIPTION:
Physical fitness is one of the leading concepts of health and well-being at all stages of life. In certain context, individuals tend to engage in prolonged sedentary behaviors, and these contexts are considered sedentary-promoting environments. These environments also detrimental on physical fitness and health. University students and office workers who predominantly engage in sedentary behaviors, such as prolonged sitting and computer-based work, have consistently shown associations with various aspects of diminished physical fitness. The online intervention protocols might be a good alternative for increasing fitness level for those who live or work in highly sedentary settings. Hence, the purpose of this study is to investigate the effectiveness of 8-week online delivered exercise program on actual and perceived physical fitness components. Specifically, body composition measured by DXA, upper body muscular strength, and flexibility are the main focus of this study. Moreover, physical self-perception is also a focus of this study.

ELIGIBILITY:
Inclusion Criteria:

* Working or studying at the university,
* Do not have any health problems that would prevent from participating in exercise,
* Not participating any another exercise/training program during the research process,
* Voluntarily participation
* Being suitable for exercise participation according to Physical Activity Readiness Questionnaire (PARQ) test results

Exclusion Criteria:

* Presence of any significant health conditions that may pose a risk during exercise (e.g., heart conditions, severe respiratory disorders, uncontrolled hypertension).
* A history of musculoskeletal injuries or conditions that would limit participation in physical fitness activities.
* Current or recent participation in another exercise or fitness program.
* Inability to provide informed consent or unwillingness to participate voluntarily.
* Any medical condition that contraindicates exercise or physical activity as determined by a healthcare professional.
* Pregnancy or postpartum period, depending on the specific requirements and goals of the intervention.
* Age restrictions (younger than 18).
* Cognitive impairments that would hinder the ability to understand and follow exercise instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Total Fat Mass | 8 weeks
  Body fat mass is the weight of fat in the body, and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Fat Mass in Legs | 8 weeks
  Fat mass in legs is the weight of fat in legs, and measured by Dual-Energy X-Ray.Absorptiometry (DXA). The unit of measurement is expressed in grams
Fat Mass in Arms | 8 weeks
  Fat mass in arms is the weight of fats in arms, and measured by Dual-Energy X-Ray Absorptiometry (DXA).The unit of measurement is expressed in grams
Fat Mass in Trunk | 8 weeks
  Fat mass in trunk is the weight of fats in trunk and measured by Dual-Energy X-Ray Absorptiometry (DXA).The unit of measurement is expressed in grams
Fat Mass in Gynoid | 8 weeks
  The Gynoid region is that around the hips and thighs. Fat mass in gynoid is the weight of fats in gynoid region and measured by Dual-Energy X-Ray Absorptiometry (DXA).The unit of measurement is expressed in grams
Fat Mass in Android | 8 weeks
  The Android region is that of the abdomen, Fat mass in android region is the weight of fats in this region and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Total Muscle Mass | 8 weeks
  Total muscle mass is the weight of muscle in the body and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Muscle Mass in Legs | 8 weeks
  Muscle mass in legs is the weight of muscle in the leg region and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Muscle Mass in Arms | 8 weeks
  Muscle mass in arms is the weight of muscle in arms and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Muscle Mass inTrunk | 8 weeks
  Muscle mass in trunk is the weight of muscle in trunk region and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Muscle Mass in Android | 8 weeks
  The Android region is that of the abdomen; muscle mass in android is the weight of muscle in android region and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams
Muscle Mass in Gynoid | 8 weeks
  The Gynoid region is that around the hips and thighs; muscle mass in gynoid is the weight of muscle in gynoid region and measured by Dual-Energy X-Ray Absorptiometry (DXA). The unit of measurement is expressed in grams

SECONDARY OUTCOMES:
Push-Up Test | 2 months
  Participants were asked to place their hands flat on the ground under their shoulders, with a straight slanted line on shoulders, back and legs. While performing the test, participants were expected to lowered the torso until the elbows are in line until 90 degrees angle with upper arms and shoulders were parallel to the ground, while the body were lifted up until the arms are straight at the lifting part. Participants were asked to perform push-ups every 3 seconds and an auditory stimulus was utilized, they were instructed to do each repetition with their body moving rigidly in a roughly straight line.
Curl-Up Test | 8 weeks
  The participants were told to lay supine on a mat with the knees bent at a 90 degrees angle, the legs spread apart, and the arms completely extended at the sides with the middle finger of both hands contacting a piece of tape. The zero point was marked with the first piece of tape, and a second piece was placed 10 cm away. A metronome was set to 20 repetitions per minute. In time with the metronome, the participant was directed to curl up until his middle finger reached the second piece of tape.
Sit and Reach Test | 8 weeks
  A sit and reach box (Lafayette Instrument Company, USA) with a scale marked on the upper side were placed against the wall. The participants were seated barefoot, with their legs fully extended and hip-width apart from the testing box. Participants were instructed to slowly reach forward and slide their fingers along the scale on top of the box by placing one hand over the other. The goal was for participants to maintain the position for about 3 seconds with their knees as straight as they could The final position that the participant reaches were recorded to the nearest centimeter and set as the score for the test.
Perceived Body Fat | 8 weeks
  Perceived body fat is one's own assessment of his or her own body fat. The body fat subscale of Marsh's Physical Self-Description Questionnaire (PSDQ) was used to collect physical self-perception data. The subscale consisted of six items, answered on a 7-point Likert scale. The maximum score that can be obtained from this scale is 42, and the minimum score is 6. The higher scores obtained in the subdimensions represent higher physical self-perception.
Perceived Physical Strength | 8 weeks
  Perceived physical strength is one's own assessment of his or her own strength. The strength subscale of Marsh's Physical Self-Description Questionnaire (PSDQ) was used to collect physical self-perception data. The subscale consisted of six items, answered on a 7-point Likert scale. The maximum score that can be obtained from this scale is 42, and the minimum score is 6. The higher scores obtained in the subdimensions represent higher physical self-perception.
Perceived Flexibility | 8 weeks
  Perceived flexibility is one's own assessment of his or her own flexibility. The flexibility subscale of Marsh's Physical Self-Description Questionnaire (PSDQ) was used to collect physical self-perception data. The subscale consisted of six items, answered on a 7-point Likert scale. The maximum score that can be obtained from this scale is 42, and the minimum score is 6. The higher scores obtained in the subdimensions represent higher physical self-perception.
Perceived Physical Health | 8 weeks
  Perceived physical health is one's own assessment of his or her own health. The physical health subscale of Marsh's Physical Self-Description Questionnaire (PSDQ) was used to collect physical self-perception data. The subscale consisted of eight items, answered on a 7-point Likert scale. The maximum score that can be obtained from this scale is 42, and the minimum score is 8. The higher scores obtained in the subdimensions represent higher physical self-perception.

CONTACTS AND LOCATIONS:
Overall Officials: Günay Yıldızer, Ph.D., Principal Investigator — Eskişehir Tech. Uni.
Locations (1):
- Eskişehir Technical University, Eskişehir, Tepebaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No